CLINICAL TRIAL: NCT01151033
Title: A Clinical Evaluation of the ProNOVA XR Polymer Free Drug Eluting Coronary Stent System in the Treatment of Patients With de Novo Coronary Artery Lesions
Brief Title: A Clinical Evaluation of the ProNOVA XR Polymer Free Drug Eluting Coronary Stent System
Acronym: EURONOVA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: KCRI (Other)
Collaborators: Vascular Concepts Limited (Industry)
Responsible Party: Swaminathan Jayaraman, CEO, Vascular Concepts Limited
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XR I
Record Dates: First submitted 2010-06-18; First posted 2010-06-25 (Estimated); Last update posted 2011-01-20 (Estimated); Status verified 2011-01

CONDITIONS: Myocardial Ischemia
Keywords: ProNOVA XR Polymer Free Drug Eluting Coronary Stent System; DES; stent; coronary artery lesions; ProNOVA; stent implantation
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- stent implantation (Experimental): ProNOVA XR Polymer Free Drug Eluting Stent implantation - single arm
  Interventions: Device: Drug Eluting Stent implantation

INTERVENTIONS:
Device: Drug Eluting Stent implantation — ProNOVA XR Drug Eluting Stent implantation

SUMMARY:
The objective of this study is the assessment of the performance, safety and efficacy of the ProNOVA XR Polymer Free Drug Eluting Stent System in the treatment of patients with de novo native coronary artery lesions.

DETAILED DESCRIPTION:
This study is a prospective, single arm, multicenter registry of approximately 50 patients undergoing PCI with the ProNOVA Drug Eluting Coronary Stent System according to its Instructions for Use.

The purpose of this registry is the evaluation of the performance, safety and efficacy of ProNOVA XR DES in real-world patients. Following initial stent implantation, all patients will have clinical follow up at 30 days, at 6 and 12 months. Additionally all patients will have a angiographic F/U at 6 months to assess the late luminal loss by QCA measurements and the neointimal volume including stent apposition by intravascular ultrasound.

ELIGIBILITY:
General Inclusion Criteria:

* Patient must be at least 18 years of age.
* Patient is able to verbally confirm understanding of risks, benefits and treatment alternatives of receiving the ProNOVA XR DES and she or her legally authorized representative provides written informed consent prior to any study related procedure, as approved by the appropriate Medical Ethics Committee of the respective clinical site.
* Patient must have evidence of myocardial ischemia (e.g., stable or unstable angina, silent ischemia, positive functional study or a reversible change in the electrocardiogram (ECG) consistent with ischemia)
* Patient must agree to undergo all required follow-up examinations.
* Patients of childbearing potential must have had a negative pregnancy test within 7 days before treatment, and must not be nursing at the time of treatment.

Angiographic Inclusion Criteria:

* Target lesions must be de novo lesions (no prior stent implant, no prior brachytherapy)
* Target vessel reference diameter must be between 2.25 mm and 4.0 mm by visual estimate
* Target lesion ≤ 28 mm in length by visual estimate

Exclusion Criteria:

* Patient has other medical illness (e.g., cancer or congestive heart failure) or known history of substance abuse (alcohol, cocaine, heroin etc.) that may cause non-compliance with the clinical investigation plan, confound the data interpretation or is associated with a limited life expectancy (i.e., less than one year)
* Patient has a known hypersensitivity or contraindication to aspirin, either heparin or bivalirudin, both clopidogrel and ticlopidine, cobalt, chromium, nickel, or contrast sensitivity that cannot be adequately pre-medicated
* Participation in another device or drug study or has completed the follow-up phase of another study within the last 30 days
* Patients judged to have a lesion that prevents complete inflation of an angioplasty balloon.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
In-stent late luminal loss | at 6 months after stent implantation

SECONDARY OUTCOMES:
Clinically and non-clinically indicated target lesion revascularization | at 30 days
Clinically and non-clinically indicated target vessel revascularization | at 30 days
Incidence of total and cardiovascular death | at 30 days
Incidence of nonfatal myocardial infarction | at 30 days
Definite, probable, and possible stent thrombosis | at 30 days
Clinically and non-clinically indicated target lesion revascularization | at 6 months
Clinically and non-clinically indicated target vessel revascularization | at 6 months
Incidence of total and cardiovascular death | at 6 months
Incidence of nonfatal myocardial infarction | at 6 months
Definite, probable, and possible stent thrombosis | at 6 months
Clinically and non-clinically indicated target lesion revascularization | at 12 months
Clinically and non-clinically indicated target vessel revascularization | at 12 months
Incidence of total and cardiovascular death | at 12 months
Incidence of nonfatal myocardial infarction | at 12 months
Definite, probable, and possible stent thrombosis | at 12 months
In-stent and in-segment percent diameter stenosis (% DS) | at 6 months after stent implantation
In-stent and in-segment binary restenosis rate as assessed by QCA | at 6 months after stent implantation
In-stent and in-segment minimal luminal diameter (MLD)as assessed by QCA | at 6 months after stent implantation
In-stent and in-segment late luminal loss as assessed by QCA | at 6 months after stent implantation
Neointimal hyperplasia as assessed by intravascular ultrasound (IVUS) | at 6 months after stent implantation
Rate of incomplete stent apposition as assessed by intravascular ultrasound (IVUS) | at 6 months after stent implantation

CONTACTS AND LOCATIONS:
Overall Officials: Dariusz Dudek, MD, PhD, Principal Investigator — Department of Haemodynamics and Angiocardiography Medical College Jagiellonian University University Hospital in Krakow
Locations (3):
- Poland (3):
  - Department of Haemodynamics and Angiocardiography Medical College Jagiellonian University University Hospital in Krakow, Krakow
  - Oddział Kardiologii Inwazyjnej Elektroterapii i Angiologii NZOZ Nowy Sacz, Nowy Sącz
  - Oddział Kardiologii Inwazyjnej Elektroterapii i Angiologii NZOZ Nowy Targ, Nowy Targ